CLINICAL TRIAL: NCT00981474
Title: Continuous Cerebral Autoregulation Monitoring to Reduce Brain Injury From Cardiac Surgery
Brief Title: Cerebral Autoregulation Monitoring During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Charles W Hogue, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 680; 1R01HL092259 (NIH)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-01

CONDITIONS: Thoracic Surgery; Cardiopulmonary Bypass
Keywords: cardiac surgery; brain injury; cerebral autoregulation
MeSH Terms: conditions — Brain Injuries | interventions — Homeostasis; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Blood pressure targets during cardiopulmonary bypass based on institutional standards of empiric management.
  Interventions: Device: Control group
- Intervention (Experimental): Blood pressure management based on cerebral autoregulation data.
  Interventions: Drug: blood pressure maintenance based on cerebral blood flow autoregulation measurement

INTERVENTIONS:
Drug: blood pressure maintenance based on cerebral blood flow autoregulation measurement — Blood pressure lowered or raised
  Other Names: Autoregulation
  Arms: Intervention
Device: Control group — Institutional standard of care.
  Other Names: Usual (Control Group)
  Arms: Control

SUMMARY:
Neurological complications from cardiac surgery are an important source of operative mortality, prolonged hospitalization, health care expenditure, and impaired quality of life. New strategies of care are needed to avoid rising complications for the growing number of aged patients undergoing cardiac surgery. This study will evaluate novel methods for reducing brain injury during surgery from inadequate brain blood flow using techniques that could be widely employed.

DETAILED DESCRIPTION:
Brain injury during cardiac surgery results primarily from cerebral embolism and/or reduced cerebral blood flow (CBF). The latter is of particular concern for the growing number of surgical patients who are aged and/or who have cerebral vascular disease. Normally, CBF is physiologically autoregulated (or kept constant) within a range of blood pressures allowing for stable cerebral O2 supply commensurate with metabolic demands. Cerebral autoregulation is impaired in patients undergoing cardiac surgery who have cerebral vascular disease and in many others due to other conditions. This could lead to brain injury since current practices of targeting low mean arterial blood pressure empirically (usually 50-70 mmHg) during cardiopulmonary bypass may expose patients with impaired cerebral autoregulation to cerebral hypoperfusion. The hypothesis of this proposal is that targeting mean arterial pressure during cardiopulmonary bypass to a level above an individual's lower autoregulatory threshold reduces the risk for brain injury in patients undergoing cardiac surgery. Monitoring of cerebral autoregulation will be performed in real time using software that continuously compares the relation between arterial blood pressure and CBF velocity of the middle cerebral artery measured with transcranial Doppler and with cerebral oximetry measured with near infrared spectroscopy. The primary end-point of the study will be a comprehensive composite outcome of clinical stroke, cognitive decline, and/or new ischemic brain lesions detected with diffusion weighted magnetic resonance (MR) imaging. Delirium assessed using a validated procedure that includes validated tools is a secondary outcome measure. Autoregulation is mediated by reactivity of cerebral resistance vessels. A secondary aim of this proposal is to evaluate whether near infrared reflectance spectroscopy can be used to trend changes in cerebral blood volume and provide a reliable monitor of vascular reactivity (the hemoglobin volume index). Assessments for extra-cranial and intra-cranial arterial stenosis will be performed using MR angiography to control for this potential confounding variable in the analysis. Finally, an additional aim of the study will be to assess whether preoperative transcranial Doppler examination of major cerebral arteries can identify patients who are prone to the composite neurological end-point. Near infrared oximetry is non-invasive, continuous, requires little care-giver intervention and, thus, could be widely used to individualize patient blood pressure management during surgery. Brain injury from cardiac surgery is an important source of operative mortality, prolonged hospitalization, increased health care expenditure, and impaired quality of life. Developing strategies to reduce the burden of this complication has wide public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients undergoing primary or re-operative Coronary Artery Bypass Graft (CABG) and/or valvular surgery or ascending aorta surgery that requires Cardio-pulmonary bypass (CPB) who are at high risk for neurologic complications (stroke or encephalopathy) as determined by a Johns Hopkins risk score of >0.02

Exclusion Criteria:

* Contraindication to MRI imaging (e.g., permanent pacemaker, cerebral arterial vascular clips)
* Liver function test before surgery more than twice the upper limit of institutional normal
* Pre-existing renal dysfunction defined as an estimated glomerular filtration rate of ≤60 mL/min, or current renal dialysis
* Emergency surgery
* Inability to attend outpatient visits
* Visual impairment or inability to speak and read English. The patient will be excluded from further study if an adequate temporal window for Transcranial Doppler (TCD) monitoring can not be identified before surgery.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hogue, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hogue CW Jr, Palin CA, Arrowsmith JE. Cardiopulmonary bypass management and neurologic outcomes: an evidence-based appraisal of current practices. Anesth Analg. 2006 Jul;103(1):21-37. doi: 10.1213/01.ANE.0000220035.82989.79. PMID 16790619
- [Background] Gottesman RF, Hillis AE, Grega MA, Borowicz LM Jr, Selnes OA, Baumgartner WA, McKhann GM. Early postoperative cognitive dysfunction and blood pressure during coronary artery bypass graft operation. Arch Neurol. 2007 Aug;64(8):1111-4. doi: 10.1001/archneur.64.8.noc70028. Epub 2007 Jun 11. PMID 17562924
- [Background] Gottesman RF, Sherman PM, Grega MA, Yousem DM, Borowicz LM Jr, Selnes OA, Baumgartner WA, McKhann GM. Watershed strokes after cardiac surgery: diagnosis, etiology, and outcome. Stroke. 2006 Sep;37(9):2306-11. doi: 10.1161/01.STR.0000236024.68020.3a. Epub 2006 Jul 20. PMID 16857947
- [Background] Nomura Y, Faegle R, Hori D, Al-Qamari A, Nemeth AJ, Gottesman R, Yenokyan G, Brown C, Hogue CW. Cerebral Small Vessel, But Not Large Vessel Disease, Is Associated With Impaired Cerebral Autoregulation During Cardiopulmonary Bypass: A Retrospective Cohort Study. Anesth Analg. 2018 Dec;127(6):1314-1322. doi: 10.1213/ANE.0000000000003384. PMID 29677060
- [Background] Czosnyka M, Brady K, Reinhard M, Smielewski P, Steiner LA. Monitoring of cerebrovascular autoregulation: facts, myths, and missing links. Neurocrit Care. 2009;10(3):373-86. doi: 10.1007/s12028-008-9175-7. Epub 2009 Jan 6. PMID 19127448
- [Background] Brady K, Joshi B, Zweifel C, Smielewski P, Czosnyka M, Easley RB, Hogue CW Jr. Real-time continuous monitoring of cerebral blood flow autoregulation using near-infrared spectroscopy in patients undergoing cardiopulmonary bypass. Stroke. 2010 Sep;41(9):1951-6. doi: 10.1161/STROKEAHA.109.575159. Epub 2010 Jul 22. PMID 20651274
- [Background] Piechnik SK, Yang X, Czosnyka M, Smielewski P, Fletcher SH, Jones AL, Pickard JD. The continuous assessment of cerebrovascular reactivity: a validation of the method in healthy volunteers. Anesth Analg. 1999 Oct;89(4):944-9. doi: 10.1097/00000539-199910000-00023. PMID 10512269
- [Background] Kneebone AC, Andrew MJ, Baker RA, Knight JL. Neuropsychologic changes after coronary artery bypass grafting: use of reliable change indices. Ann Thorac Surg. 1998 May;65(5):1320-5. doi: 10.1016/s0003-4975(98)00158-1. PMID 9594860
- [Background] Brown CH 4th, Probert J, Healy R, Parish M, Nomura Y, Yamaguchi A, Tian J, Zehr K, Mandal K, Kamath V, Neufeld KJ, Hogue CW. Cognitive Decline after Delirium in Patients Undergoing Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):406-416. doi: 10.1097/ALN.0000000000002253. PMID 29771710
- [Background] Brown CH 4th, Neufeld KJ, Tian J, Probert J, LaFlam A, Max L, Hori D, Nomura Y, Mandal K, Brady K, Hogue CW; Cerebral Autoregulation Study Group; Shah A, Zehr K, Cameron D, Conte J, Bienvenu OJ, Gottesman R, Yamaguchi A, Kraut M. Effect of Targeting Mean Arterial Pressure During Cardiopulmonary Bypass by Monitoring Cerebral Autoregulation on Postsurgical Delirium Among Older Patients: A Nested Randomized Clinical Trial. JAMA Surg. 2019 Sep 1;154(9):819-826. doi: 10.1001/jamasurg.2019.1163. PMID 31116358
- [Background] Goldstein LB, Bertels C, Davis JN. Interrater reliability of the NIH stroke scale. Arch Neurol. 1989 Jun;46(6):660-2. doi: 10.1001/archneur.1989.00520420080026. PMID 2730378
- [Background] Evered L, Eckenhoff RG; International Perioperative Cognition Nomenclature Working Group. Perioperative cognitive disorders. Response to: Postoperative delirium portends descent to dementia. Br J Anaesth. 2017 Dec 1;119(6):1241. doi: 10.1093/bja/aex404. No abstract available. PMID 29156035
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Lameire N, Kellum JA; KDIGO AKI Guideline Work Group. Contrast-induced acute kidney injury and renal support for acute kidney injury: a KDIGO summary (Part 2). Crit Care. 2013 Feb 4;17(1):205. doi: 10.1186/cc11455. PMID 23394215
- [Background] Mathew JP, Mackensen GB, Phillips-Bute B, Grocott HP, Glower DD, Laskowitz DT, Blumenthal JA, Newman MF; Neurologic Outcome Research Group (NORG) of the Duke Heart Center. Randomized, double-blinded, placebo controlled study of neuroprotection with lidocaine in cardiac surgery. Stroke. 2009 Mar;40(3):880-7. doi: 10.1161/STROKEAHA.108.531236. Epub 2009 Jan 22. PMID 19164788
- [Background] Vedel AG, Holmgaard F, Rasmussen LS, Langkilde A, Paulson OB, Lange T, Thomsen C, Olsen PS, Ravn HB, Nilsson JC. High-Target Versus Low-Target Blood Pressure Management During Cardiopulmonary Bypass to Prevent Cerebral Injury in Cardiac Surgery Patients: A Randomized Controlled Trial. Circulation. 2018 Apr 24;137(17):1770-1780. doi: 10.1161/CIRCULATIONAHA.117.030308. Epub 2018 Jan 16. PMID 29339351
- [Background] Gold JP, Charlson ME, Williams-Russo P, Szatrowski TP, Peterson JC, Pirraglia PA, Hartman GS, Yao FS, Hollenberg JP, Barbut D, et al. Improvement of outcomes after coronary artery bypass. A randomized trial comparing intraoperative high versus low mean arterial pressure. J Thorac Cardiovasc Surg. 1995 Nov;110(5):1302-11; discussion 1311-4. doi: 10.1016/S0022-5223(95)70053-6. PMID 7475182
- [Background] Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, Beyersdorf F. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011 Jul;40(1):200-7. doi: 10.1016/j.ejcts.2010.11.024. Epub 2010 Dec 18. PMID 21168339
- [Background] Joshi B, Ono M, Brown C, Brady K, Easley RB, Yenokyan G, Gottesman RF, Hogue CW. Predicting the limits of cerebral autoregulation during cardiopulmonary bypass. Anesth Analg. 2012 Mar;114(3):503-10. doi: 10.1213/ANE.0b013e31823d292a. Epub 2011 Nov 21. PMID 22104067
- [Background] Cook DJ, Huston J 3rd, Trenerry MR, Brown RD Jr, Zehr KJ, Sundt TM 3rd. Postcardiac surgical cognitive impairment in the aged using diffusion-weighted magnetic resonance imaging. Ann Thorac Surg. 2007 Apr;83(4):1389-95. doi: 10.1016/j.athoracsur.2006.11.089. PMID 17383345
- [Background] Vedel AG, Holmgaard F, Siersma V, Langkilde A, Paulson OB, Ravn HB, Nilsson JC, Rasmussen LS. Domain-specific cognitive dysfunction after cardiac surgery. A secondary analysis of a randomized trial. Acta Anaesthesiol Scand. 2019 Jul;63(6):730-738. doi: 10.1111/aas.13343. Epub 2019 Mar 19. PMID 30891734
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Brown CH 4th, Laflam A, Max L, Lymar D, Neufeld KJ, Tian J, Shah AS, Whitman GJ, Hogue CW. The Impact of Delirium After Cardiac Surgical Procedures on Postoperative Resource Use. Ann Thorac Surg. 2016 May;101(5):1663-9. doi: 10.1016/j.athoracsur.2015.12.074. Epub 2016 Mar 31. PMID 27041454
- [Background] Gottesman RF, Grega MA, Bailey MM, Pham LD, Zeger SL, Baumgartner WA, Selnes OA, McKhann GM. Delirium after coronary artery bypass graft surgery and late mortality. Ann Neurol. 2010 Mar;67(3):338-44. doi: 10.1002/ana.21899. PMID 20373345
- [Background] Brady KM, Lee JK, Kibler KK, Smielewski P, Czosnyka M, Easley RB, Koehler RC, Shaffner DH. Continuous time-domain analysis of cerebrovascular autoregulation using near-infrared spectroscopy. Stroke. 2007 Oct;38(10):2818-25. doi: 10.1161/STROKEAHA.107.485706. Epub 2007 Aug 30. PMID 17761921
- [Derived] Lewis C, Dokucu ME, Brown CH, Balmert L, Srdanovic N, Madhan AS, Samra SS, Csernansky J, Grafman J, Hogue CW. Postoperative but not preoperative depression is associated with cognitive impairment after cardiac surgery: exploratory analysis of data from a randomized trial. BMC Anesthesiol. 2022 May 23;22(1):157. doi: 10.1186/s12871-022-01672-y. PMID 35606688
- [Derived] Nakano M, Nomura Y, Suffredini G, Bush B, Tian J, Yamaguchi A, Walston J, Hasan R, Mandal K, Schena S, Hogue CW, Brown CH 4th. Functional Outcomes of Frail Patients After Cardiac Surgery: An Observational Study. Anesth Analg. 2020 Jun;130(6):1534-1544. doi: 10.1213/ANE.0000000000004786. PMID 32384343
- [Derived] Nomura Y, Nakano M, Bush B, Tian J, Yamaguchi A, Walston J, Hasan R, Zehr K, Mandal K, LaFlam A, Neufeld KJ, Kamath V, Hogue CW, Brown CH 4th. Observational Study Examining the Association of Baseline Frailty and Postcardiac Surgery Delirium and Cognitive Change. Anesth Analg. 2019 Aug;129(2):507-514. doi: 10.1213/ANE.0000000000003967. PMID 30540612
- [Derived] Hori D, Katz NM, Fine DM, Ono M, Barodka VM, Lester LC, Yenokyan G, Hogue CW. Defining oliguria during cardiopulmonary bypass and its relationship with cardiac surgery-associated acute kidney injury. Br J Anaesth. 2016 Dec;117(6):733-740. doi: 10.1093/bja/aew340. PMID 27956671
- [Derived] Brown CH 4th, Faigle R, Klinker L, Bahouth M, Max L, LaFlam A, Neufeld KJ, Mandal K, Gottesman RF, Hogue CW Jr. The Association of Brain MRI Characteristics and Postoperative Delirium in Cardiac Surgery Patients. Clin Ther. 2015 Dec 1;37(12):2686-2699.e9. doi: 10.1016/j.clinthera.2015.10.021. Epub 2015 Nov 29. PMID 26621626
- [Derived] Hori D, Brown C, Ono M, Rappold T, Sieber F, Gottschalk A, Neufeld KJ, Gottesman R, Adachi H, Hogue CW. Arterial pressure above the upper cerebral autoregulation limit during cardiopulmonary bypass is associated with postoperative delirium. Br J Anaesth. 2014 Dec;113(6):1009-17. doi: 10.1093/bja/aeu319. Epub 2014 Sep 25. PMID 25256545
- [Derived] Ono M, Brady K, Easley RB, Brown C, Kraut M, Gottesman RF, Hogue CW Jr. Duration and magnitude of blood pressure below cerebral autoregulation threshold during cardiopulmonary bypass is associated with major morbidity and operative mortality. J Thorac Cardiovasc Surg. 2014 Jan;147(1):483-9. doi: 10.1016/j.jtcvs.2013.07.069. Epub 2013 Sep 26. PMID 24075467

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining written informed consent, 468 were randomized to the two groups. 237 in the autoregulation group were randomized after consent and 5 subjects withdrew consent. 231 in the usual care group were randomized after consent and 3 subjects withdrew consent.
Groups:
- Usual Care Group (Control): Blood pressure targets during cardiopulmonary bypass based on institutional standards of empiric management.
  Control group: Institutional standard of care.
- Autoregulation Group: Blood pressure management based on cerebral autoregulation data.
  blood pressure maintenance based on cerebral blood flow autoregulation measurement: Blood pressure lowered or raised
Period: Overall Study
Arm/Group | Usual Care Group (Control) | Autoregulation Group
Started | 228 | 232
Completed | 228 | 232
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Group: Blood pressure targets during cardiopulmonary bypass based on institutional standards of empiric management.
  Control group: Institutional standard of care.
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Autoregulation Group | Total
Number analyzed (Participants) | 228 | 232 | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.0) | 70.0 (7.3) | 70.4 (7.6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 67 | 62 | 129
  Male | 160 | 170 | 330
  Missing designation | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 189 | 184 | 273
  African American | 24 | 28 | 52
  Hispanic | 3 | 2 | 5
  Native American | 1 | 3 | 4
  Asian | 0 | 4 | 4
  Multiple | 0 | 2 | 2
  Other | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 228 | 232 | 460
Highest Grade of Formal Education (median,[inter-quartile range]) [Median (Inter-Quartile Range); unit: Years] | 14.0 [12 to 17] | 14.5 [12 to 17] | 14 [12 to 17]
Mini-Mental State Exam [Median (Inter-Quartile Range); unit: score on a scale (30 good- 0 poor)] — The Mini-Mental Status Examination tests for quantify cognitive function and screens for cognitive loss. It assesses the individual's orientation, attention, calculation, recall, language and motor skills. The highest score (no deficits, good ) is 30 and a score under 20 suggests a mental deficit (poor).
  score on a scale (30 good- 0 poor) | 28 [27 to 29] | 28 [26 to 29] | 28 [26 to 29]
History of a prior stroke [Count of Participants; unit: Participants] | 25 | 19 | 44
History of hypertension [Count of Participants; unit: Participants] | 213 | 207 | 420
History of atrial fibrillation [Count of Participants; unit: Participants] | 53 | 49 | 102
History of myocardial infarction [Count of Participants; unit: Participants] | 65 | 74 | 139
History of chronic obstructive lung disease [Count of Participants; unit: Participants] | 31 | 21 | 52
Obstructive sleep apnea [Count of Participants; unit: Participants] | 41 | 36 | 77
Current tobacco use [Count of Participants; unit: Participants] | 22 | 24 | 46
History of diabetes [Count of Participants; unit: Participants] | 101 | 108 | 209
History of anemia [Count of Participants; unit: Participants] | 101 | 108 | 209
Logistic EuroSCORE (median,[interquartile range]) [Median (Inter-Quartile Range); unit: score on a scale 0-2 good >=5 high risk] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) identifies a number of risk factors which help to predict mortality from cardiac surgery. the predicted mortality (in percent) is calculated by adding the weights assigned to each risk factor.It comprises 18 variables, weighted from 1-4, and defines low risk as 0-2 points (0.8% mortality), medium risk as 3-5 points (3.0% mortality), and high risk as > 5 points (11% mortality).
  score on a scale 0-2 good >=5 high risk | 5.3 [2.99 to 10.97] | 5.08 [2.56 to 11.62] | 5.19 [2.56 to 11.62]
Cardiopulmonary bypass duration [Median (Inter-Quartile Range); unit: Minutes] | 107 [81.5 to 140.5] | 103 [81 to 141] | 105 [81 to 141]
Type of surgery [Count of Participants; unit: Participants]
  Coronary Artery Bypass Graft (CABG) | 109 | 117 | 226
  Coronary Aertery Bypass Graft, Aortic Valve Replacement (CABG/AVR) | 35 | 26 | 61
  Coronary Artery Bypass Graft, Mitral Valve Replacement CABG/MVR) | 6 | 9 | 15
  Coronary Artery Bypass Graft, Aortic Valve Replacement, Mitral Valve Replacement (CABG/AVR/MVR) | 3 | 3 | 6
  Aortic Valve Replacement (AVR) | 41 | 48 | 89
  Mitral Valve Replacement (MVR) | 19 | 22 | 41
  Aortic Valve Replacement, Mitral Valve Replacement (AVR/MVR) | 9 | 5 | 14
  Aortic Root Replacement | 2 | 2 | 4
  Coronary Artery Bypass Graft, (CABG) / Aortic Root Replacement | 1 | 0 | 1
  Transcatheter Aortic Valve Replacement (TAVR) | 3 | 0 | 3
Aortic cross-clamp (time in minutes) [Median (Inter-Quartile Range); unit: Minutes] | 73 [53 to 93.5] | 69 [54 to 93.25] | 71 [53 to 93.25]
Duration of ICU admission (hours) [Median (Inter-Quartile Range); unit: Hours] | 44.1 [27.1 to 86.1] | 44 [24 to 68.7] | 44 [24 to 86.1]
Duration of hospitalization (days) [Median (Inter-Quartile Range); unit: Days] | 8 [6 to 11] | 7 [6 to 10] | 7 [6 to 11]
Cardiopulmonary bypass duration [Median (Inter-Quartile Range); unit: Minutes] | 107 [81.5 to 140.5] | 103 [81 to 141] | 105 [81 to 141]

OUTCOME MEASURES:

1. Primary Outcome: Composite Neurological Outcome of Clinical Stroke or New Ischemic Brain Lesion on Diffusion Weighted MRI or Neurocognitive Dysfunction 4 to 6 Weeks After Surgery.
Description: The composite neurological outcome was composed of clinical stroke, or new ischemic lesions detected on postoperative brain diffusion weighted magnetic resonance imaging(DWI), or cognitive decline from baseline to 4-6 weeks after surgery.
Time Frame: Up to 6 weeks post-operative
Population: Subjects who completed neurological testing and MRI testing
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (Control) | Autoregulation Group
Number analyzed (Participants) | 101 | 93
Participants | 79 | 70
Statistical Analysis 1: Comparison: Usual Care Group (Control) vs Autoregulation Group; Test type: Superiority; p = .752, Chi-squared; Risk Ratio (RR) = .96, 95% CI 2-sided [.82 to 1.121]

2. Secondary Outcome: Postoperative Delirium
Description: Assessed with Confusion Assessment Method or Confusion Assessment Method-ICU along with adjudication by team of experts
Time Frame: Postoperative days 1-4
Population: Delirium was measured day 1-4. 232 in the autoregulation group were assessed and 228 were assessed in the usual care group.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group (Control) | Autoregulation Group
Number analyzed (Participants) | 228 | 232
Participants | 34 | 19
Statistical Analysis 1: Comparison: Usual Care Group (Control) vs Autoregulation Group; Test type: Superiority; p = .053, Chi-squared; Risk Ratio (RR) = .55, 95% CI 2-sided [.32 to .93]

3. Secondary Outcome: Multiple Inotropic Drugs>24 Hours After Surgery
Description: Use of multiple inotropic drugs greater than 24 hours after the planned surgical procedure until discharge from the hospital.
Time Frame: 7 days after surgery
Population: 228 in the usual care group and 232 in the autoregulation group were analyzed.
Measure: Number; unit: participants
Arm/Group | Usual Care Group (Control) | Autoregulation Group
Number analyzed (Participants) | 228 | 232
participants | 13 | 6
Statistical Analysis 1: Comparison: Usual Care Group (Control) vs Autoregulation Group; Test type: Superiority; p = .149, Chi-squared; Risk Ratio (RR) = .454, 95% CI 2-sided [.18 to 1.17]

4. Secondary Outcome: Mechanical Lung Ventilation>24 Hours After Surgery
Description: Subjects need for mechanical lung ventilation more than 24 hours after planned surgical procedure.
Time Frame: Up to 28 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 22 | 13
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .144, Chi-squared; Hazard Ratio (HR) = .581, 95% CI 2-sided [.30 to 1.13]

5. Secondary Outcome: Insertion of Intra-aortic Balloon Pump
Description: Procedural insertion of intra-aortic balloon pump within 7 days after surgical procedure
Time Frame: 7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 19 | 14
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .439, Chi-squared; Risk Ratio (RR) = .724, 95% CI 2-sided [.37 to 1.41]

6. Secondary Outcome: Postoperative Atrial Fibrillation
Description: Clinical diagnosis of postoperative atrial fibrillation from date of surgical procedure to discharge from the hospital.
Time Frame: Up to 28 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 89 | 79
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .311, Chi-squared; Risk Ratio (RR) = .872, 95% CI 2-sided [.69 to 1.11]

7. Secondary Outcome: Sepsis
Description: Clinical diagnosis of sepsis from time of surgical procedure to discharge from the hospital.
Time Frame: Up to 28 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 7 | 2
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .103, Fisher Exact; Fisher exact test used due to the small number of events; Risk Ratio (RR) = .247, 95% CI 2-sided [.005 to 1.18]

8. Secondary Outcome: Acute Kidney Injury Within 7 Days After Surgery.
Description: Subject developed acute kidney injury within 7 days after surgical procedure. Based on Kidney disease: Improving Global Outcomes (KDIGO) classification system.
Time Frame: 7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 56 | 62
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .608, Chi-squared; Risk Ratio (RR) = 1.102, 95% CI 2-sided [.81 to 1.5]

9. Secondary Outcome: New Renal Replacement Therapy
Description: Subjects requiring new renal replacement therapy prior to discharge from hospital
Time Frame: Up to 28 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 6 | 4
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .541, Fisher Exact; Fisher exact test used due to the small number of events; Risk Ratio (RR) = .564, 95% CI 2-sided [.16 to 1.97]

10. Secondary Outcome: Multisystem Organ Failure After Surgery
Description: Subject diagnosis of multisystem organ failure after surgery.
Time Frame: Up to 28 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 7 | 2
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .103, Fisher Exact; Fisher exact test used due to small number of events; Risk Ratio (RR) = .247, 95% CI 2-sided [.05 to 1.18]

11. Secondary Outcome: Mortality
Description: Subject death within 28 days after surgical procedure
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 228 | 232
Participants | 12 | 5
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .129, Chi-squared; Risk Ratio (RR) = .409, 95% CI 2-sided [.15 to 1.14]

ADVERSE EVENTS:
Time Frame: Data were collected over a period of 1 year.
Description: Postoperative complications were based on the Society of Thoracic Surgery National Cardiac Surgery Database definitions (www.sts.org) as safety outcomes.
Arm/Group | Usual Care Group (Control) | Autoregulation Group
All-Cause Mortality (participants affected / at risk) | 12/228 | 5/232
Serious Adverse Events (participants affected / at risk) | 133/228 | 121/232
Other Adverse Events (participants affected / at risk) | 34/228 | 19/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Usual Care Group (Control) (N=228) | Autoregulation Group (N=232)
Acute Kidney Injury (Renal and urinary disorders) | 56 (56) | 62 (62) — Acute kidney injury within 7 days after surgical procedure. Based on Kidney Disease: Improving Global Outcomes (KDIGO) classification system.
Multisystem Organ Failure after Surgery (General disorders) | 6 (6) | 4 (4)
Sepsis (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Clinical Stroke (Nervous system disorders) | 9 (9) | 13 (13)
New Ischemic Lesions in Brian (Nervous system disorders) | 47/85 (47) | 48/79 (48) — New ischemic lesions detected on subjects who completed postoperative brain diffusion weighted magnetic resonance imaging (DWI)
Delayed Neurocognitive Recovery (General disorders) | 35/164 (35) | 27/172 (27) — Of the number of subjects who completed the neurocognitive testing in the post operative period.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (Control) (N=228) | Autoregulation Group (N=232)
Clinically detected delirium (Psychiatric disorders) | 34 (34) | 19 (19) — Clinically detected delirium by the caregivers in the hospital setting. Post-operative day 1 to day of discharge.

LIMITATIONS AND CAVEATS:
Limitations include missing data including unavoidable missing MRI data (retained temporary cardiac pacemaker leads, patient refusal and discharge prior to scheduled MRI. Patient refusal of completing cognitive tests. Enrollment period of 9 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT00981474/Prot_SAP_000.pdf